CLINICAL TRIAL: NCT07232719
Title: A Phase 3b Study to Investigate the Efficacy and Safety of Retatrutide Once Weekly in Participants Without Type 2 Diabetes Who Have Obesity or Overweight: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Study of Retatrutide (LY3437943) in Participants With Obesity or Overweight
Acronym: TRIUMPH-8
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27769; J1I-MC-GZQJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — retatrutide

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide subcutaneously (SC)
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide SC
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of retatrutide compared with placebo for body weight reduction.

Participation in the study will last about 65 weeks and may include about 18 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of:

  * ≥30 kilogram per square meter (kg/m2) OR
  * ≥27 kg/m2 with at least one of the following weight-related conditions: high blood pressure, abnormal levels of lipid, obstructive sleep apnea, heart disease
* Have at least one unsuccessful attempt to lose weight by dieting

Exclusion Criteria:

* Have a self-reported change in body weight >5 kg (11 pounds) within 90 days before screening
* Have a prior or planned surgical treatment for obesity
* Have type 1 diabetes or type 2 diabetes
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had within the past 90 days before screening

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * hospitalization for unstable angina, or
  * hospitalization due to congestive heart failure
* Have New York Heart Association Functional Classification Class IV congestive heart failure
* Have a history of chronic or acute pancreatitis
* Have taken weight loss drugs, including over-the counter medications within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 56

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure | Baseline, Week 56
Change from Baseline in Waist Circumference | Baseline, Week 56
Percent Change from Baseline in Non-High-Density Lipoprotein (HDL) Cholesterol | Baseline, Week 56
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) | Baseline through Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (19):
  - Artemis Institute for Clinical Research, Riverside, California
  - JEM Research Institute, Atlantis, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - Care Access - Arlington Heights, Arlington Heights, Illinois
  - L-MARC Research Center, Louisville, Kentucky
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - IMA Clinical Research Manhattan, New York, New York
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Cedar Health Research, Dallas, Texas
  - Headlands Research-El Paso, El Paso, Texas
  - Cedar Health Research - Euless, Euless, Texas
  - Cedar Health Research - Fort Worth, Fort Worth, Texas
  - Care Access - Houston, Houston, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
- United Kingdom (12):
  - FutureMeds - Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - FutureMeds - Liverpool, Bromborough
  - Cheadle Community Hospital, Cheadle
  - HMC Health Group - Meadows Centre for Health, Hounslow
  - St Bartholomew's Medical Centre, Oxford
  - Atlantic Medical, Penzance
  - The Adam Practice, Poole
  - Woodstock Bower Surgery, Rotherham
  - Rame Group Practice, Torpoint
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants with Obesity or Overweight (TRIUMPH-8) — https://trials.lilly.com/en-US/trial/667856